CLINICAL TRIAL: NCT02095158
Title: A Long-term Safety and Efficacy Study of Oxymetazoline HCl Cream 1.0% in Patients With Persistent Erythema Associated With Rosacea
Brief Title: A Long-Term Safety and Efficacy Study AGN-19920 in Patients With Persistent Erythema Associated With Rosacea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 199201-006
Record Dates: First submitted 2014-03-21; First posted 2014-03-24 (Estimated); Results first posted 2016-09-21 (Estimated); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Erythema; Rosacea
MeSH Terms: conditions — Erythema; Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxymetazoline HCL Cream 1.0% (Experimental): Oxymetazoline HCL Cream 1.0% (AGN-199201) applied to the face once daily for 52 weeks.
  Interventions: Drug: Oxymetazoline HCL Cream 1.0%

INTERVENTIONS:
Drug: Oxymetazoline HCL Cream 1.0% — Oxymetazoline HCL Cream 1.0% applied to the face once daily for 52 weeks.
  Other Names: AGN-199201

SUMMARY:
This study will evaluate the long-term safety and efficacy of oxymetazoline hydrogen chloride (HCL) Cream 1.0% (AGN-199201) in patients with persistent erythema associated with rosacea.

ELIGIBILITY:
Inclusion Criteria:

-Moderate to severe persistent facial erythema associated with rosacea.

Exclusion Criteria:

* Current treatment with monoamine oxidase (MAO) inhibitors
* Raynaud's syndrome, narrow angle glaucoma, orthostatic hypotension, scleroderma or Sjogren's syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxymetazoline HCL Cream 1.0%: Oxymetazoline hydrogen chloride (HCL) Cream 1.0% (AGN-199201) applied to the face once daily for 52 weeks.
Period: Overall Study
Arm/Group | Oxymetazoline HCL Cream 1.0%
Started | 440
Completed | 365
Not Completed | 75
Not completed — Adverse Event | 14
Not completed — Lack of Efficacy | 3
Not completed — Pregnancy | 1
Not completed — Lost to Follow-up | 20
Not completed — Personal Reasons | 35
Not completed — Protocol Violation | 1
Not completed — Other Miscellaneous Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxymetazoline HCL Cream 1.0%
Number analyzed (Participants) | 440
Age, Customized [Number; unit: participants]
  18 to 64 years | 370
  ≥ 65 years | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 335
  Male | 105

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Related Adverse Events
Description: An adverse event was considered any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug. A Treatment-Related Adverse Event is an Adverse Event determined by the investigator to be causally related to the study medication.
Time Frame: 56 Weeks
Population: Safety population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | Oxymetazoline HCL Cream 1.0%
Number analyzed (Participants) | 440
percentage of participants | 8.2

2. Secondary Outcome: Percentage of Participants With at Least a 2-Grade Decrease From Baseline on Both Clinician Erythema Assessment (CEA) and Subject Satisfaction Assessment (SSA) Using 5-Point Scales
Description: The investigator assessed the participant's overall severity of erythema in the treatment area by using the 5-point CEA scale with photonumeric guide where: 0=clear skin with no signs of erythema (best) to 4=severe erythema; fiery redness (worst). A decrease in the score indicates improvement. The participant assessed their overall severity of rosacea facial redness in the treatment area by using the 5-point SSA scale with photoguide where: 0=no signs of unwanted redness (best) to 4=severe redness (worst). A decrease in the score indicates improvement. The percentage of participants with at least a 2-grade decrease (improvement) on both CEA and SSA from Baseline was evaluated over the 6-hour evaluation period (hours 3 and 6) post-dose.
Time Frame: Baseline, Day 1 Hours 3 and 6, Week 4 Predose and Hours 3 and 6, Week 12 Predose, Week 26 Predose and Hours 3 and 6, Week 39 Predose, Week 52 Predose and Hours 3 and 6, Week 54 Predose
Population: Modified-intent-to-treat (mITT) population consisted of all participants who had at least 1 post-baseline CEA and SSA measurement.
Measure: Number; unit: percentage of participants
Arm/Group | Oxymetazoline HCL Cream 1.0%
Number analyzed (Participants) | 440
percentage of participants
  Day 1 (Hour 3) | 11.6
  Day 1 (Hour 6) | 17.8
  Week 4 (Predose) | 1.2
  Week 4 (Hour 3) | 19.5
  Week 4 (Hour 6) | 23.0
  Week 12 (Predose) | 6.1
  Week 26 (Predose) | 6.5
  Week 26 (Hour 3) | 34.7
  Week 26 (Hour 6) | 38.1
  Week 39 (Predose) | 9.5
  Week 52 (Predose) | 11.2
  Week 52 (Hour 3) | 36.7
  Week 52 (Hour 6) | 43.4
  Week 54 (Predose) | 12.1

ADVERSE EVENTS:
Time Frame: Up to 56 Weeks
Arm/Group | Oxymetazoline HCL Cream 1.0%
Serious Adverse Events (participants affected / at risk) | 15/440
Other Adverse Events (participants affected / at risk) | 0/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxymetazoline HCL Cream 1.0% (N=440)
Angina pectoris (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Chest pain (General disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Appendicitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Chronic sinusitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parkinson's disease (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.